CLINICAL TRIAL: NCT00773240
Title: A Phase III Trial Assessing the Pharmacodynamic Effect and the Tolerability of Grazax Treatment Initiated in the Grass Pollen Season in Subjects With Seasonal Grass Pollen Induced Rhinoconjunctivitis
Brief Title: A Phase III Trial Assessing the Pharmacodynamic Effect and the Tolerability of Grazax Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GT-18
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Grass Pollen Allergy
MeSH Terms: interventions — Grazax

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Grazax
  Interventions: Drug: Grazax
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Grazax — 1 tablet, 75,000 SQ-T, daily during the trial period
  Arms: 1
Drug: placebo — 1 placebo tablet, matching the active treatment, daily during the trial period
  Arms: 2

SUMMARY:
The study assess the pharmacodynamic effect and the tolerability of Grazax treatment initiated in the grass pollen season in subjects with seasonal grass pollen induced rhinoconjunctivitis

ELIGIBILITY:
Inclusion Criteria:

* Positive skin prick test to Phleum pratense
* Positive IgE to Phleum pratense
* signed informed consent
* A clinical history of moderate to severe persistent rhinoconjunctivitis symptoms

Exclusion Criteria:

* No uncontrolled asthma in the past 12 months
* No history of an IgE mediated systemic reaction due to food, insect venom, any kind of medication or induced by exercise, where there are symptoms both from the skin and the respiratory system with or without hypotension
* No history of an IgE mediated systemic reaction due to food, insect venom, any kind of medication or induced by exercise, where there are symptoms both from the skin and the respiratory system with or without hypotension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2008-04; Primary Completion 2008-10 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics - Immunological assessments | Pre- and post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kim Simonsen, MD, Study Director — ALK-Abelló A/S
Locations (1):
- ALK-Abello A/S, Bøge alle 6-8, Hørsholm, Denmark

REFERENCES:
- [Derived] Reich K, Gessner C, Kroker A, Schwab JA, Pohl W, Villesen H, Wustenberg E, Emminger W. Immunologic effects and tolerability profile of in-season initiation of a standardized-quality grass allergy immunotherapy tablet: a phase III, multicenter, randomized, double-blind, placebo-controlled trial in adults with grass pollen-induced rhinoconjunctivitis. Clin Ther. 2011 Jul;33(7):828-40. doi: 10.1016/j.clinthera.2011.06.006. Epub 2011 Jul 7. PMID 21741092